CLINICAL TRIAL: NCT01742026
Title: ADVANCE THERAPY ASPERGILLOSIS INVASIVE IN PATIENTS HIGH RISK ONCOHEMATOLOGICAL PCR USING FOR EARLY DETECTION OF ASPERGILLUS
Brief Title: Aspergillus PCR Early Detection in High Risk Oncohematological Patients
Acronym: PCRAGA
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Other Study IDs: GETH-PCRAGA
Record Dates: First submitted 2012-10-30; First posted 2012-12-05 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Infections
Keywords: High risk aspergillosis infection patients
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High Risk Oncohematological Patients: Detection Aspergillus PCR technique and Aspergillus AGA technique
  Interventions: Procedure: Aspergillus PCR technique; Procedure: Aspergillus AGA technique

INTERVENTIONS:
Procedure: Aspergillus PCR technique — Aspergillus DNA PCR technique
Procedure: Aspergillus AGA technique — Aspergillus AGA technique

SUMMARY:
ADVANCE THERAPY ASPERGILLOSIS INVASIVE BY PCR DETECTION

DETAILED DESCRIPTION:
ADVANCE THERAPY ASPERGILLOSIS INVASIVE IN PATIENTS HIGH RISK ONCOHEMATOLOGICAL PCR USING FOR EARLY DETECTION OF ASPERGILLUS

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent to participate in the study.
* Adult patients (> 18 years), diagnosed with acute myelogenous leukemia or myelodysplastic syndrome with chemotherapy (CT) intensive, or admitted to undergo allogeneic hematopoietic progenitor cells, or transplantation with graft versus host disease.
* The patient should be included in this protocol from the start of their chemotherapy or conditioning therapy as reflected in another section.

Exclusion Criteria:

* Employment of antifungal prophylaxis (30 days prior to inclusion) with triazole / polyene with activity against Aspergillus (itraconazole, voriconazole, posaconazole, amphotericin B inhalation).
* Use of other systemic antifungal activity against Aspergillus (amphotericin, terbinafine, flucytosine, echinocandins, etc.). Therefore it will Fluconazole prophylaxis exclusively.
* Background of IFI proven / probable prior
* Probable IFI / tested at the time of inclusion in the study.
* Exclusion will cause a lack of compliance with the inclusion criteria.
* Patients who have a lack of follow biweekly with galactomannan or PCR. Have a bacterial infection not properly treated and controlled before starting empirical antifungal treatment (according to the definition given above). And finally they have a neutropenia of short duration that it creates a significant risk of IFI. This information will not be known logically to include the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of hematological patients at high risk of invasive fungal infection. Like: Leukemia acute mieloblasticas, myelodysplastic syndrome, patients with intensive chemotherapy and allogeneic hematopoietic transplantation.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of PCR technique for detection of Aspergillus DNA versus the standard technique for the determination of galactomannan Antigen (AGA) in serum | 18-20 months
  To value the percentage of patients with likely/proven invasive fungal infection, diagnosed using only AGA tecnique or using AGA and PCR tecniques together.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Vazquez, MD, Principal Investigator — University of Salamanca; Isabel Ruiz, Md, Principal Investigator — Hospital Vall d´Hebron; Rocio Parody, MD, Principal Investigator — Hospital Virgen del Rocio; Javier Lopez, MD, Principal Investigator — Hospital Ramon y Cajal; Montserrat Rovira, MD, Principal Investigator — Hospital Clinic of Barcelona; Montserrat Batlle, MD, Principal Investigator — Germans Trias i Pujol Hospital; Carlos Vallejo, MD, Principal Investigator — Hospital Central de Asturias; Rosario Varela, MD, Principal Investigator — Hospital de A Coruña; Inmaculada Heras, MD, Principal Investigator — Hospital Morales Meseguer; Joaquin Diaz, MD, Principal Investigator — Hospital Clinico San Carlos; Carlos Solano, MD, Principal Investigator — Hospital Clinico de Valencia; Maria Teresa Olave, MD, Principal Investigator — Hospital Lozano Blesa; David Gallardo, MD, Principal Investigator — H. Josep Trueta
Locations (13):
- Spain (13):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario de A Coruña, A Coruña
  - Hospital Vall d´Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital morales Meseguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Virgen del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Aguado JM, Vazquez L, Fernandez-Ruiz M, Villaescusa T, Ruiz-Camps I, Barba P, Silva JT, Batlle M, Solano C, Gallardo D, Heras I, Polo M, Varela R, Vallejo C, Olave T, Lopez-Jimenez J, Rovira M, Parody R, Cuenca-Estrella M; PCRAGA Study Group; Spanish Stem Cell Transplantation Group; Study Group of Medical Mycology of the Spanish Society of Clinical Microbiology and Infectious Diseases; Spanish Network for Research in Infectious Diseases. Serum galactomannan versus a combination of galactomannan and polymerase chain reaction-based Aspergillus DNA detection for early therapy of invasive aspergillosis in high-risk hematological patients: a randomized controlled trial. Clin Infect Dis. 2015 Feb 1;60(3):405-14. doi: 10.1093/cid/ciu833. Epub 2014 Oct 21. PMID 25336623